CLINICAL TRIAL: NCT00109759
Title: A Double-Blind Phase I Study to Evaluate the Safety and Tolerability of Tyrosine Adsorbed Ragweed Pollen Allergoid With MPL® in Healthy Volunteers.
Brief Title: Evaluation of Safety and Tolerability of Tyrosine Adsorbed Ragweed Pollen Allergoid With MPL (Monophosphoryl Lipid A)
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Allergy Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RagweedMATAMPL102; P1DP05002
Record Dates: First submitted 2005-05-03; First posted 2005-05-04 (Estimated); Last update posted 2021-08-12 (Actual); Status verified 2021-07

CONDITIONS: Type I Hypersensitivity
Keywords: allergy; allergoid; specific immunotherapy; ragweed; Tyrosine
MeSH Terms: conditions — Hypersensitivity, Immediate; Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- RagweedMATAMPL (Experimental)
  Interventions: Biological: RagweedMATAMPL
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: RagweedMATAMPL
  Arms: RagweedMATAMPL
Drug: Placebo
  Arms: Placebo

SUMMARY:
The safety and tolerability of tyrosine adsorbed ragweed pollen allergoid with monophosphoryl lipid A (MPL) was planned to be evaluated. For this purpose, a total of 4 injections of either increasing doses of the study drug or placebo (tyrosine) was planned to be administered in 7-day intervals to healthy volunteers.

DETAILED DESCRIPTION:
RagweedMATAMPL (tyrosine adsorbed ragweed pollen allergoid with monophosphoryl lipid A (MPL®)) has been developed to provide pre-seasonal specific immunotherapy for patients with proven type I hypersensitivity to ragweed pollen. MPL (Monophosphoryl Lipid A), a purified, detoxified glycolipid derived from the cell wall of Salmonella minnesota, is included in the product formulation as an adjuvant to increase the immunogenic effect of the product and to enhance the switch from an allergen-specific TH2 to a TH1-like profile.

The ragweed pollen extract is modified with glutaraldehyde to produce the active ingredient, an allergoid. This modification reduces the reactivity of the extract with IgE antibody, thus reducing the risk of side effects. However, a simultaneous reduction in other important immunological properties, such as IgG and T cell reactivities is not seen.

This was planned to be a phase I, double-blind, placebo-controlled study to evaluate the safety and tolerability of RagweedMATAMPL in healthy volunteers. Fifteen (15) volunteers were planned to be randomized to receive up to 4 subcutaneous injections of either increasing doses of RagweedMATAMPL or Placebo over 7 day intervals.

ELIGIBILITY:
Inclusion Criteria:

* Non-smoker and not using any nicotine products
* Negative skin prick test with a standard panel of marker allergen extracts (including ragweed allergen extract)
* Specific IgE for ragweed with class = 0
* No clinical history of IgE-mediated allergic diseases
* Subject agrees not to use any medication or herbal products during the study
* Males or non-pregnant, non-lactating females who are post-menopausal, naturally or surgically sterile, or who agree to use effective contraceptive methods throughout the course of the study.
* Subjects who are normally active and otherwise judged to be in good health on the basis of medical history, physical examination, routine laboratory tests and an infection screen
* Subjects must be willing and able to attend required study visits.
* Subjects must be able to follow instructions.

Exclusion Criteria:

* Clinical history or presence of acute or subacute atopic dermatitis, chronic dermatitis, urticaria factitia, or urticaria due to physical/chemical influence.
* Clinical history or presence of diabetes, cancer or any clinically significant cardiac, respiratory, metabolic, renal, hepatic, gastrointestinal, dermatologic, venereal, hematologic, neurologic or psychiatric diseases or disorders.
* Any clinically significant (as determined by the Investigator) abnormal laboratory value at Visit 1
* Clinical history of auto-immune diseases or rheumatoid diseases.
* Contraindication to adrenaline
* History of asthma
* Subject has used any prescription medications within 14 days or over-the-counter medications, including herbal products, within 2 days prior to Screening or will likely use any medication(s) or listed product(s) during the study.
* Subject has disorder of tyrosine metabolism
* Subject with diseases with a pathogenesis interfering with the immune response and who has received medication which could influence the results of this study
* Subject has acute or chronic infection
* Clinical history of anaphylaxis
* Clinical history of angioedema
* Clinical history of hypersensitivity to the excipients of the study medication
* History of immunotherapy with ragweed allergen extracts
* Current therapy with ß-blockers
* Currently receiving anti-allergy medication or other drugs with an antihistaminic activity
* Subject has a positive screen for cotinine or drugs of abuse at Visit 1
* Subject has a positive saliva alcohol test at Visit 1
* Subject participated in a clinical trial with a new chemical substance within the last 12 months
* Subject cannot communicate reliably with the Investigator or is not likely to cooperate with the requirements of the study
* Subject is pregnant or lactating
* Clinically relevant abnormal vital signs or respiratory rate at the Screening Visit
* Subject received treatment with a preparation containing MPL® during the past 12 months.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2005-05; Study Completion 2005-06

PRIMARY OUTCOMES:
Safety and tolerability | 29 days
  Recording of adverse events (AEs).

SECONDARY OUTCOMES:
Tolerability of different subcutaneous doses | 29 days
  Recording of adverse events (AEs).
Tolerability of the cumulative subcutaneous dose | 29 days
  Recording of adverse events (AEs).
Clinical chemistry, hematology, respiratory rate, and ECG before and after each dose and at the end of the study | 29 days

CONTACTS AND LOCATIONS:
Locations (1):
- Allied Research International Inc., Mississauga, Ontario, Canada